CLINICAL TRIAL: NCT06024356
Title: Efficacy and Safety of Neoadjuvant Chemoradiotherapy Combined With PD-1 Inhibitor and Thymalfasin for Locally Advanced Mid-low Rectal Cancer: a Single-center, Retrospective, Controlled Study
Brief Title: Neoadjuvant Chemoradiotherapy Combined With PD-1 Inhibitor and Thymalfasin for Locally Advanced Mid-low Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Other Study IDs: BFH-TTNCRT
Record Dates: First submitted 2023-08-08; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Programmed Cell Death 1 Receptor; Thymalfasin; Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Thymalfasin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Pathology Paraffin Sections （Pre-NCRT and Post-NCRT）
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: long course radiotherapy (50 Gy/25f, 2 Gy/f, 5 days/week) for the first 5 weeks and three 21-day cycles capecitabine (1000 mg/m2, bid, po, day1-14) plus three 21-day cycles tislelizumab (200 mg, iv.gtt, day 8) for the first 9 weeks. After that, patients rested for two weeks (week 10-11)。6-8 weeks after the end of radiotherapy, patients underwent TME surgery (12-14 weeks). Thymalfasin was started on the first day of neoadjuvant chemoradiotherapy, 1.6 mg subcutaneously twice a week until the end of the last neoadjuvant treatment.
  Interventions: Drug: Thymalfasin
- Control: long course radiotherapy (50 Gy/25f, 2 Gy/f, 5 days/week) for the first 5 weeks and three 21-day cycles capecitabine (1000 mg/m2, bid, po, day1-14) plus three 21-day cycles tislelizumab (200 mg, iv.gtt, day 8) for the first 9 weeks. After that, patients rested for two weeks (week 10-11)。6-8 weeks after the end of radiotherapy, patients underwent TME surgery (12-14 weeks).

INTERVENTIONS:
Drug: Thymalfasin — Thymalfasin (thymosin-alpha 1) is an immunomodulating agent able to enhance the Thl immune response. It has been evaluated for its immunomodulatory activities and related therapeutic potential in several diseases.
  Groups: Experimental

SUMMARY:
It is a single-center, retrospective, controlled study to investigate the efficacy and safety of neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and thymalfasin for locally advanced mid-low rectal cancer.

DETAILED DESCRIPTION:
Study Purpose

1. To evaluate the efficacy and safety of neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and thymalfasin for locally advanced mid-low rectal cancer.
2. To explore the effects of neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and thymalfasin on the immune microenvironment of locally advanced mid-low rectal cancer.

Study Design: A single-center, retrospective, controlled study Subjects were divided into two groups according to whether or not they received thymalfasin: group 1 was treated with neoadjuvant chemoradiotherapy combined with PD-1 inhibitor, and group 2 was treated with neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and thymalfasin.

Subjects received long course radiotherapy (50 Gy/25f, 2 Gy/f, 5 days/week) for the first 5 weeks and three 21-day cycles capecitabine (1000 mg/m2, bid, po, day1-14) plus three 21-day cycles tislelizumab (200 mg, iv.gtt, day 8) for the first 9 weeks. After that, patients rested for two weeks (week 10-11)。6-8 weeks after the end of radiotherapy, patients underwent TME surgery (12-14 weeks). Thymalfasin was started on the first day of neoadjuvant chemoradiotherapy, 1.6 mg subcutaneously twice a week until the end of the last neoadjuvant treatment.

Enrollment: 26 participants, 13 in each group Study Population: locally advanced mid-low rectal cancer Primary Endpoint: pathologic complete response（pCR） Exploratory endpoint: Paraffin specimens were collected from biopsies before neoadjuvant therapy and after surgery in patients meeting the inclusion criteria. The expression of CD86, CD163, CD4+T，CD8+T，PD-1 were detected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal adenocarcinoma must satisfied all the following conditions:

  1. Stage II/III LARC (cT1-4aN0-2M0);
  2. Tumor distal location≤10 cm from anal verge (MRI diagnosed);
* Patients regardless of gender with aged≥18 years
* ECOG score of 0 or 1
* Physical and viscera function of patients can withstand major abdominal surgery

Exclusion Criteria:

* Current or previous active malignancy other than rectal cancer；
* Patients underwent major surgery within 4 weeks prior to neoadjuvant therapy；
* Patients have any condition affects the absorption of capecitabine through gastrointestinal tract；
* Patients have severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
* Patients with severe concomitant diseases with estimated survival≤5 years；
* Patients with present or previous moderate or severe liver and kidney damage；
* Patients preparing for or previously received organ or bone marrow transplant；
* Patients who have received immunosuppressive or systemic hormone therapy within 1 month prior to the start of neoadjuvant therapy；
* Patients with congenital or acquired immune deficiency (such as HIV infection)；
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced mid-low rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | 1 year
  All the enrolled patients will receive total mesorectal excision (TME) 7-9 weeks after the end of long course radiotherapy. The rectal specimens will be evaluated by the pathologists who are experienced on the rectal cancer diagnosis according to the 1997 Dworak grading system. The rectal cancer will be classified into 5 grades. Grade 0-3 will be considered as non-pCR while grade 4 represent pCR.

SECONDARY OUTCOMES:
neoadjuvant rectal (NAR) score | 1 year
  The neoadjuvant rectal (NAR) score is a promising indicator of survival after preoperative chemoradiotherapy for rectal cancer. The NAR score was calculated according to the following formula: NAR score = [5pN - 3(cT - pT) + 12]2⁄9.61.
  (clinical tumor (cT) stage, pathologic tumor (pT) stage, pathologic nodal (pN) stage)
tumor regression grade（TRG） | 1 year
  AJCC 8th TRG classification. TRG 0: No viable cancer cells left in the specimen; complete regression.
  TRG 1: Minimal residual cancer cells present; extensive regression with a minimal number of tumor cells.
  TRG 2: Moderate residual cancer cells present; substantial regression with a significant number of tumor cells.
  TRG 3: Minimal or no regression; no significant tumor cell response to treatment; majority of tumor still present.
objective response rate (ORR) | 1 year
  ORR is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The ORR rate is the sum of complete response (CR) and partial response (PR)
R0 resection rate | 1 year
  During the surgical process, the surgeon will evaluate the level of cancer resection. It will be classified as R0, R1, R2 resection. Therefore, we can calculate R0 resection rate.
anal preservation rate | 1 year
  the surgeon will decide whether the anal can be preserved on the basis of the rectal cancer and intraoperative situation. anal preservation rate is the percentage of patients who achieve anal preservation.
disease free survival (DFS) | 3 year
  During the 3-year follow-up, the percentage of the patients who is disease free.
local recurrence free survival | 3 year
  During the 3-year follow-up, the percentage of local recurrence.
overall survival (OS) | 3 year
  During the 3-year follow-up, the percentage of the patients who is sill survival at the end of follow-up.

OTHER OUTCOMES:
The expression of CD86 | 1 year
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD163 | 1 year
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD4+ | 1 year
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD8+ | 1 year
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of PD-1 | 1 year
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital medical University, Beijing, Xicheng Dis, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025.5-
Access Criteria: via reasonable email requests